CLINICAL TRIAL: NCT01283620
Title: Atlantic Canada Modified Constraint Induced Movement Therapy Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Dalhousie University (Other); Sunnybrook Research Institute (Other)
Responsible Party: Principal Investigator, Shaun Boe, Affiliate Scientist, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDHA-RS/2011-277
Record Dates: First submitted 2011-01-21; First posted 2011-01-26 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Stroke
Keywords: stroke; extremity, upper
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Other)
  Interventions: Other: Usual and Customary Care
- modified CIMT (mCIMT) (Experimental)
  Interventions: Behavioral: modified constraint induced movement therapy (mCIMT)

INTERVENTIONS:
Behavioral: modified constraint induced movement therapy (mCIMT) — The intervention group will receive usual care plus mCIMT. mCIMT consists of two components delivered in parallel: three 30 min therapy sessions/week focusing on progressively more difficult tasks performed with the arm/hand, and five hours/weekday of restraint of the unaffected upper limb. Each 30 min therapy session consists of using the affected upper limb in practicing 4-5 functionally relevant tasks.
  Arms: modified CIMT (mCIMT)
Other: Usual and Customary Care — Patients in this arm will receive usual care dose-matched to the experimental care group. Usual care will consist of occupational and physiotherapy intervention focused on affected upper limb range of motion (i.e., active range of motion incorporated into functional tasks such as reaching), strengthening (i.e., upper limb resisted exercise), manual dexterity exercises (i.e., grasp and release, stacking cones), and general aerobic conditioning (i.e., recumbent stepper, treadmill).
  Arms: Usual Care

SUMMARY:
The purpose of this study is to examine the effectiveness and feasibility of a modified constraint induced movement therapy (mCIMT) intervention on upper limb function in two groups of patients acutely post-stroke; 1) an experimental group that will participate in a 10 week mCIMT intervention designed to improve upper limb function, in addition to usual care, and 2) a control group that will participate in a program of usual care consisting of a rehabilitation intervention for the affected upper limb that is dose-matched to the experimental group.

ELIGIBILITY:
Inclusion Criteria:

1. first symptomatic stroke (either ischemic or hemorrhagic) resulting in upper limb hemiparesis
2. the ability to perform a two-step command
3. age ≥ 18 years
4. residence within a 75 km radius of the Queen Elizabeth II Health Sciences Centre
5. with regard to the affected upper limb, subjects will meet standard criteria for modified constraint induced movement therapy (mCIMT) including at least 10 degrees of active wrist extension, at least 10 degrees of thumb abduction/extension, and at least 10 degrees of extension in two additional digits, repeated three times in one minute

Exclusion Criteria:

1. have excessive pain in the affected upper limb (defined as > 4 on a 10 centimeter visual analog scale)
2. presence of dementia or aphasia as defined by a score of < 26 on the Montreal Cognitive Assessment
3. have a diagnosis of pre-stroke dementia
4. have a terminal illness, life-threatening co-morbidity or concomitant neurological or psychiatric illness
5. excessive tone in the upper limb (> 3 on the modified Ashworth Scale)
6. Motor Activity Log score > 2.5 (amount of use sub-scale)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in arm and hand function at 10 weeks, 6 and 12 months relative to baseline performance | At 0 weeks, 10 weeks, 6 months and 12 months
  Change in arm and hand function will be performed using the Action Research Arm Test, which measures function of the arm and hand using 19 tasks in four different categories (grip, grasp, pinch and gross motor). Performance on each task is scored from 0 (cannot perform any part of the test) to 3 (performs the test normally) for a possible score of 0-57. Improved arm and hand function will be determined by detecting a change in score by comparing performance at each of the post-treatment assessment points (10 weeks, 6 and 12 months) relative to baseline performance.

SECONDARY OUTCOMES:
Change in the quality and amount of arm and hand use at 10 weeks, 6 and 12 months relative to baseline. | At 0 weeks, 10 weeks, 6 months and 12 months
  Improved arm and hand function based on the quality and amount of use will be determined by detecting a change in score by comparing performance at each post-treatment assessment point (10 weeks, 6 and 12 months) relative to baseline performance using the Motor Activity Log. The Motor Activity Log is a semi-structured interview which measures how much and how well a person is using the affected arm and hand compared to their pre-stroke condition.
Greater satisfaction with treatment compared to the usual care group based on higher scores on the Satisfaction with Stroke Care Questionnaire (SASC-19) in the experimental treatment group | At 10 weeks
  Overall satisfaction with treatment will be measured in each group using the Satisfaction with Stroke Care Questionnaire (SASC-19), which includes 19 questions relating to a patients satisfaction with their care and treatment.
Improved return to normal activities in the experimental treatment group as measured by higher scores on the Re-integration to Normal Living Index (RNLI) 6 months post-treatment | At 6 months
Change in the amount of use of the arm and hand in everyday life at 10 weeks, 6 and 12 months relative to baseline as detected with accelerometers | At 0 weeks, 10 weeks, 6 months and 12 months
  Accelerometers will be worn on both wrists to quantitatively assess the amount of movement that occurs over a three day period at each of the time points. Improved use of the arm and hand will be determined based on a change in activity at each of the post-treatment assessment points (10 weeks, 6 and 12 months) relative to activity measured at baseline.
Improved return to normal activities in the experimental treatment group as measured by higher scores on the Re-integration to Normal Living Index (RNLI) 12 months post-treatment | At 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Shaun G Boe, MPT, PhD, Principal Investigator — Dalhousie University/Capital Health
Locations (1):
- Capital Health, Halifax, Nova Scotia, Canada